CLINICAL TRIAL: NCT01824836
Title: A Cohort Study to Evaluate Genetic Predictors of Aromatase Inhibitor Musculoskeletal Symptoms (AIMSS)
Brief Title: A Study to Evaluate Genetic Predictors of Aromatase Inhibitor Musculoskeletal Symptoms (AIMSS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E1Z11; NCI-2013-00426 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA037403 (NIH)
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Results first posted 2025-04-24 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-03

CONDITIONS: Estrogen Receptor-positive Breast Cancer; Musculoskeletal Complications; Progesterone Receptor-positive Breast Cancer; Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (anastrozole) (Experimental): Patients receive anastrozole PO QD for 12 months.
  Interventions: Drug: anastrozole

INTERVENTIONS:
Drug: anastrozole — Given PO
  Other Names: Arimidex

SUMMARY:
E1Z11 is a study to determine whether certain genetic information can predict which breast cancer patients will discontinue treatment with aromatase inhibitors (AIs) due to the development of musculoskeletal symptoms (MSS). Women with stage I-III breast cancer who are prescribed the aromatase inhibitor anastrozole as treatment may join.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To validate previously identified associations between 10 specific single nucleotide polymorphisms (single nucleotide polymorphisms [SNPs]) and discontinuation of treatment with aromatase inhibitors (AIs) due to the development of musculoskeletal symptoms (MSS) among women with breast cancer.

SECONDARY OBJECTIVES:

I. To determine whether other SNPs in cytochrome P450 enzymes (CYP), glucuronosyltransferases (UGT), Vitamin D, serotonin and other receptors are associated with discontinuation of treatment due to the development of severe aromatase inhibitor-associated musculoskeletal symptoms (AIMSS).

II. To determine whether other SNPs in CYP, UGT, Vitamin D, serotonin and other receptors are associated with the development of other potential complications of AI therapy.

III. To develop a gene signature that can identify patients at risk for developing severe anastrozole-related AIMSS and other potential complications of AI therapy.

IV. To determine the epidemiology and predictors of severe AIMSS and of AI discontinuation.

V. To describe patient reported outcomes for minority patients with breast cancer treated with AIs.

VI. To assess the utility of the Patient Reported Outcomes Management Information System (PROMIS) system to collect patient reported outcomes in a cooperative group study, and validate the PROMIS Physical Function 20a form in patients with AIMSS.

VII. To develop a model that incorporates patient ratings of treatment burden, fear of recurrence and adherence behaviors to describe patient decisions to continue or discontinue anastrozole.

VIII. To collect serum samples for future testing for biomarkers of AIMSS.

OUTLINE:

Patients receive anastrozole orally (PO) once daily (QD) for 12 months.

After the completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be post-menopausal; post-menopausal will be defined as women meeting any of the following criteria:

  * >= 60 years of age; or
  * < 60 years of age and amenorrheic for >= 12 months prior to day 1 if uterus/ovaries are intact; or
  * < 60 years of age, and the last menstrual period 6-12 months prior to day 1, if intact uterus/ovaries and meets biochemical criteria for menopause (follicle-stimulating hormone [FSH] and estradiol within institutional standard for postmenopausal status); or
  * < 60 years of age, without a uterus, and meets biochemical criteria for menopause (FSH and estradiol within institutional standards for postmenopausal status); or
  * < 60 years of age and history of bilateral oophorectomy; surgery must have been completed at least 4 weeks prior to day 1; or
  * Prior radiation castration with amenorrhea for at least 6 months
* Patients must have estrogen and/or progesterone receptor positive histologically confirmed stage I-III adenocarcinoma of the breast
* Patients must have completed recommended local therapy and adjuvant chemotherapy for breast cancer
* Plan to treat with anastrozole for at least 12 months
* Eastern Cooperative Oncology Group (ECOG) performance status between 0-2
* Patients must be disease-free of other prior invasive malignancies for ≥ 5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix. Prior early stage breast cancers are also allowed as long as prior treatment did not include aromatase inhibitors.
* Patients must have worst pain rated as less than 4 out of 10 on the following question: "In the past week, how much pain have you had on a scale of 0 to 10, where 0 equals no pain and 10 means the worst pain you can imagine; " NOTE: This question regarding patient's pain should be completed within one week prior to registration; this pain item may be completed orally prior to consent up to 7 days prior to registration; it is not necessary to complete this pain item via the PROMIS website
* Patients must have adequate hepatic, hematologic and renal functioning to be able to be administered anastrozole at the discretion of the treating physician

Exclusion Criteria:

* Prior AI therapy with exemestane, letrozole, or anastrozole as adjuvant therapy or for prevention of breast cancer; prior tamoxifen as adjuvant therapy or for prevention is allowed
* Patients must not be currently taking (or have taken in the past 6 months) ongoing, daily analgesic medication for active, chronic conditions (i.e., rheumatoid arthritis, carpal tunnel syndrome, tenosynovitis, systemic lupus erythematosus, gout, fibromyalgia, or severe osteoarthritis involving the hands, wrists, hips, knees, feet or ankles); (note: patients taking daily low dose aspirin are allowed to participate in this trial)
* Prior history of deep vein thrombosis (DVT) or pulmonary embolism in the past 5 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1046 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, Principal Investigator — Eastern Cooperative Oncology Group
Locations (2):
- United States (2):
  - Eastern Cooperative Oncology Group, Boston, Massachusetts
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Background] Stearns V, Jegede OA, Chang VT, Skaar TC, Berenberg JL, Nand R, Shafqat A, Jacobs NL, Luginbuhl W, Gilman P, Benson AB 3rd, Goodman JR, Buchschacher GL Jr, Henry NL, Loprinzi CL, Flynn PJ, Mitchell EP, Fisch MJ, Sparano JA, Wagner LI. A Cohort Study to Evaluate Genetic Predictors of Aromatase Inhibitor Musculoskeletal Symptoms: Results from ECOG-ACRIN E1Z11. Clin Cancer Res. 2024 Jul 1;30(13):2709-2718. doi: 10.1158/1078-0432.CCR-23-2137. PMID 38640040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1046 patients were enrolled between June 11, 2013 and October 22, 2018.
Groups:
- Anastrozole: Patients receive anastrozole PO QD for 12 months.
Period: Overall Study
Arm/Group | Anastrozole
Started | 1046
Treated and Adverse Events Assessed | 1014
Evaluable Patients | 970
Evaluable Patients With rs2296972 SNP Data Available | 959
Evaluable Patients With Baseline HAQ Data Available | 954
Evaluable Patients With 3-month HAQ Data Available | 878
Evaluable Patients With 6-month HAQ Data Available | 809
Evaluable Patients With 9-month HAQ Data Available | 781
Evaluable Patients With 12-month HAQ Data Available | 772
Completed | 766
Not Completed | 280
Not completed — Adverse Event | 48
Not completed — Withdrawal by Subject | 63
Not completed — Other complicating disease | 116
Not completed — Disease progression | 5
Not completed — Alternative therapy | 2
Not completed — Depression | 1
Not completed — Non-compliance | 3
Not completed — Patient regained ovarian function | 3
Not completed — Lost to Follow-up | 8
Not completed — Physician Decision | 2
Not completed — Research office was closed | 3
Not completed — Relocation | 3
Not completed — Insurance-related issue | 1
Not completed — Transportation issue | 1
Not completed — Patient transferred care | 1
Not completed — Unknown reasons | 4
Not completed — Never started treatment | 16

BASELINE CHARACTERISTICS:
Population: All enrolled patients are included in this analysis.
Arm/Group | Anastrozole
Number analyzed (Participants) | 1046
Age, Continuous [Median (Full Range); unit: years] | 63 [31 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1046
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 1009
  Unknown or Not Reported | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 185
  Native Hawaiian or Other Pacific Islander | 9
  Black or African American | 199
  White | 631
  More than one race | 13
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Associations Between Pre-specified Single Nucleotide Polymorphisms (SNPs) and Discontinuation of Treatment With Aromatase Inhibitor (AI) Due to the Development of Musculoskeletal Symptoms (MSS)
Description: Patients were classified into two groups based on whether or not they discontinued treatment due to MSS within 12 months. The 10 SNPs evaluated include ESR1 (rs2234693, rs2347868, rs9340835), CYP19A1 (rs1062033, rs4646), TCL1A (rs11849538, rs2369049, rs7158782, rs7159713), and HTR2A (rs2296972).
  The associations between SNPs and discontinuation of treatment due to AIMSS are presented by odds ratios (ORs). An OR of 1 suggests no association, while an OR > 1 indicates a greater chance of treatment discontinuation in the one group compared to the reference group, and an OR < 1 suggests a lower chance.
Time Frame: Assessed at baseline and 3, 6, 9, 12 months
Population: Eligible and treated patients that have SNP data available were included in this analysis.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Anastrozole
Number analyzed (Participants) | 970
odds ratio
  SNP - rs1062033 : CYP19A1 | 0.89 [0.59 to 1.34]
  SNP - rs11849538 : TCL1A | 0.83 [0.49 to 1.41]
  SNP - rs2234693 : ESR1 | 1.07 [0.71 to 1.6]
  SNP - rs2296972 : HTR2A-AS1; HTR2A | 1.07 [0.71 to 1.61]
  SNP - rs2347868 : ESR1 | 1 [0.64 to 1.57]
  SNP - rs2369049 : TCL1A | 0.91 [0.59 to 1.4]
  SNP - rs4646 : CYP19A1 | 1.03 [0.66 to 1.61]
  SNP - rs7158782 : TCL1A | 0.91 [0.6 to 1.4]
  SNP - rs7159713 : TCL1A | 0.89 [0.58 to 1.37]
  SNP - rs9340835 : ESR1 | 1.18 [0.77 to 1.8]

2. Secondary Outcome: Associations Between Other SNPs in CYP, UGT, Vitamin D, Serotonin and Other Receptors and Discontinuation of Treatment Due to the Development of Severe AIMSS
Description: The associations between discontinuation of treatment due to AIMSS and various factors, including other SNPs in CYP, UGT, vitamin D, serotonin and other receptors are evaluated.
Time Frame: Assessed at baseline and 3, 6, 9, 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Associations Between Development of Other Potential Complications of AI Therapy and Other SNPs in CYP, UGT, Vitamin D, Serotonin and Other Receptors
Description: The associations between development of other potential complications of AI therapy and other SNPs in CYP, UGT, vitamin D, serotonin and other receptors are evaluated.
Time Frame: Assessed at baseline, and 3, 6, 9, 12 months
Reporting Status: Not Posted

4. Secondary Outcome: The Distribution of the Development of AIMSS by Genotype of the rs2296972 SNP
Description: The association between the rs2296972 SNP in the HTR2A-AS1;HTR2A gene and the development of AIMSS was evaluated. Patients were categorized into CC, AC and AA genotypes for the rs2296972 SNP.
  AIMSS was defined using two criteria, physician assessment and the Stanford Health Assessment Questionnaire (HAQ) score. Patients who developed joint pain or stiffness were encouraged not to discontinue treatment and were to be seen by their treating clinician within 2 weeks of the symptom(s). At the time of the visit, the treating clinician could make an AIMSS diagnosis based on a clinical assessment. AIMSS based on HAQ was defined as ≥0.20 mean increase in scaled HAQ score at 3, 6, 9 or 12 months from baseline.
Time Frame: Assessed at baseline, and 3, 6, 9, 12 months
Population: Eligible and treated patients with the rs2296972 SNP data available
Measure: Count of Participants; unit: Participants
Groups:
- CC Genotype: Patients with CC genotype for the rs2296972 SNP
- AC Genotype: Patients with AC genotype for the rs2296972 SNP
- AA Genotype: Patients with AA genotype for the rs2296972 SNP
Arm/Group | CC Genotype | AC Genotype | AA Genotype
Number analyzed (Participants) | 460 | 381 | 118
Participants
  Developed AIMSS | 179 | 170 | 60
  Did not develop AIMSS | 281 | 211 | 58

5. Secondary Outcome: The Distribution of Development of AIMSS by Race
Description: The association between race and the development of AIMSS was evaluated. AIMSS was defined using two criteria, physician assessment and the Stanford Health Assessment Questionnaire (HAQ) score. Patients who developed joint pain or stiffness were encouraged not to discontinue treatment and were to be seen by their treating clinician within 2 weeks of the symptom(s). At the time of the visit, the treating clinician could make an AIMSS diagnosis based on a clinical assessment. AIMSS based on HAQ was defined as ≥0.20 mean increase in scaled HAQ score at 3, 6, 9 or 12 months from baseline.
Time Frame: Assessed at baseline, and 3, 6, 9, 12 months
Population: Eligible and treated patients with SNP data available
Measure: Count of Participants; unit: Participants
Groups:
- Race: White: White women
- Race: Black: Black women
- Race: Asian: Asian women
Arm/Group | Race: White | Race: Black | Race: Asian
Number analyzed (Participants) | 600 | 181 | 189
Participants
  Developed AIMSS | 231 | 89 | 94
  Did not develop AIMSS | 369 | 92 | 95

6. Secondary Outcome: Patient Reported Outcomes (Health Assessment Questionnaire [HAQ] Pain Scores) at Baseline for Patients With Breast Cancer Treated With Aromatase Inhibitors (AIs).
Description: HAQ was administered to evaluate pain among the patients. The pain scores range between 0 and 3 with 0 indicating no pain and 3 indicating very severe pain.
Time Frame: Assessed at baseline
Population: Evaluable patients with baseline HAQ data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anastrozole
Number analyzed (Participants) | 954
score on a scale | 0.11 (0.14)

7. Secondary Outcome: Patient Reported Outcomes (Health Assessment Questionnaire [HAQ] Pain Scores) at 3 Months for Patients With Breast Cancer Treated With Aromatase Inhibitors (AIs).
Description: as for outcome 6
Time Frame: Assessed at 3 months
Population: Evaluable patients with 3-month HAQ data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anastrozole
Number analyzed (Participants) | 878
score on a scale | 0.14 (0.29)

8. Secondary Outcome: Patient Reported Outcomes (Health Assessment Questionnaire [HAQ] Pain Scores) at 6 Months for Patients With Breast Cancer Treated With Aromatase Inhibitors (AIs).
Description: as for outcome 6
Time Frame: Assessed at 6 months
Population: Evaluable patients with 6-month HAQ data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anastrozole
Number analyzed (Participants) | 809
score on a scale | 0.15 (0.29)

9. Secondary Outcome: Patient Reported Outcomes (Health Assessment Questionnaire [HAQ] Pain Scores) at 9 Months for Patients With Breast Cancer Treated With Aromatase Inhibitors (AIs).
Description: as for outcome 6
Time Frame: Assessed at 9 months
Population: Evaluable patients with 9-month HAQ data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anastrozole
Number analyzed (Participants) | 781
score on a scale | 0.17 (0.30)

10. Secondary Outcome: Patient Reported Outcomes (Health Assessment Questionnaire [HAQ] Pain Scores) at 12 Months for Patients With Breast Cancer Treated With Aromatase Inhibitors (AIs).
Description: as for outcome 6
Time Frame: Assessed at 12 months
Population: Evaluable patients with 12-month HAQ data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anastrozole
Number analyzed (Participants) | 772
score on a scale | 0.17 (0.31)

11. Secondary Outcome: To Develop a Model That Incorporates Patient Ratings of Treatment Burden, Fear of Recurrence and Adherence Behaviors to Describe Patient Decisions to Continue or Discontinue Anastrozole
Description: To develop a model that incorporates patient ratings of treatment burden, fear of recurrence and adherence behaviors to describe patient decisions to continue or discontinue anastrozole
Time Frame: Assessed at baseline, diagnosis of AIMSS, discontinuation of treatment due to AIMSS, one month after treatment discontinuation due to AIMSS, and 3, 6, 9, 12 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: To Assess the Utility of the Reported Outcomes Management Information System (PROMIS) to Collect Patient Reported Outcomes in a Cooperative Group Study, and Validate the PROMIS Physical Function 20a Form in Patients With AIMSS
Description: The NIH has developed a Web-based system for recording patient reported outcomes during clinical trials, the Patient Reported Outcomes Management Information System (PROMIS) that will enable the efficient collection of patient reported outcomes and decrease the logistical burdens on office practices for patients on clinical trials. The PROMIS Assessment Center is the web-based platform for dissemination of NIH PROMIS measures. The assessment center can be used to administer patient rated outcome instruments, monitor accrual, manage data, send reminders to patients, be used to deliver custom researcher developed content, and has numerous features that support both simple and complicated accrual designs.
Time Frame: as for outcome 11
Reporting Status: Not Posted

13. Other Pre Specified Outcome: To Collect Serum Samples for Future Testing for Biomarkers of AIMSS
Description: Serum samples will be collected for future testing for biomarkers of AIMSS
Time Frame: as for outcome 11
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed while on treatment and after the end of treatment up to 5 years
Description: Patients who received treatment were included in the analysis of adverse events. All patients enrolled on this study were included in the analysis of all-cause mortality.
Arm/Group | Anastrozole
All-Cause Mortality (participants affected / at risk) | 43/1046
Serious Adverse Events (participants affected / at risk) | 59/1014
Other Adverse Events (participants affected / at risk) | 546/1014
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole (N=1014)
Heart failure (Cardiac disorders) | 1
Fatigue (General disorders) | 2
Pain (General disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Weight gain (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 34
Arthritis (Musculoskeletal and connective tissue disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 3
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole (N=1014)
Arthralgia (Musculoskeletal and connective tissue disorders) | 459
Arthritis (Musculoskeletal and connective tissue disorders) | 188
Bone pain (Musculoskeletal and connective tissue disorders) | 130
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 93
Myalgia (Musculoskeletal and connective tissue disorders) | 188
Neck pain (Musculoskeletal and connective tissue disorders) | 68
Pain in extremity (Musculoskeletal and connective tissue disorders) | 198

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT01824836/Prot_SAP_000.pdf